CLINICAL TRIAL: NCT04114760
Title: Timely Acquirement of 12-lead Electrocardiography Using Patchy-type Wireless Device by Emergency Medical Technicians in Ambulance ; A Simulation Study
Brief Title: Timely Acquirement of 12-lead ECG Using Patchy-type Wireless Device by Emergency Medical Technician in Ambulance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-04-004
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chest Pain; Electrocardiography
Keywords: 12-lead electrocardiography; Emergency medical technician; chest pain; wireless technology; simulation study
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : defibrillator ECG to patchy-type ECG (Active Comparator): Group A subject will performing ECG examination to a mock patient in the ambulance.
  First ECG performance will be using defibrillator which contain 12-lead ECG checking function. And taking a 15 minutes wash out period. Second ECG performance after wash out period, will be using patchy-type wireless device.
  when ECG examination performance ended, survey of patchy-type wireless ECG device usability will be collect.
  Interventions: Device: defibrillator ECG
- Group B : patchy-type ECG to defibrillator ECG (Experimental): Group B subject will performing ECG examination to a mock patient in the ambulance.
  First ECG performance will be using patchy-type wireless device.
  And taking a 15 minutes wash out period. Second ECG performance after wash out period, will be using defibrillator which contain 12-lead ECG checking function.
  when ECG examination performance ended, survey of patchy-type wireless ECG device usability will be collect.
  Interventions: Device: patchy-type wireless ECG

INTERVENTIONS:
Device: patchy-type wireless ECG — This device consists of a single patchy and save the ECG result as a Potable Document Format. Also can transfer to hospital using wifi-network.
  Arms: Group B : patchy-type ECG to defibrillator ECG
Device: defibrillator ECG — This device is essential equipment in ambulance. For 12-lead ECG examination the connector need to replace for specific cable.
  Arms: Group A : defibrillator ECG to patchy-type ECG

SUMMARY:
In this study, the investigators compare timely acquirement and effectiveness of 12-lead ECG using patchy-type wireless versus using defibrillator which contain ECG examination function in ambulance.

The purpose of this study is to determine the difference of timely acquirement of 12-lead ECG using two different systems and the difference of efficiency of ECG examination in ambulance between two groups.

The participants in this simulation study were divided randomly into 2 groups :

Group A is performing an ECG examination on mock patient using defibrillator which contained 12-lead ECG checking function. And take a 15 minutes wash out period. After the wash out period, group A subject performing an ECG examination using patchy-type wireless device.

Group B subject is performing an ECG examination on mock patient using patchy-type wireless device first, and take a 15 minutes wash out period. After the wash out period, group B performing an ECG examination using defibrillator which contain 12-lead ECG function.

Both group's ECG examination is performing in the ambulance.

ELIGIBILITY:
Inclusion Criteria:

* Who have a certification of Emergency Medical Technician in korea and have a nurse license in korea.
* who currently engaged of emergency medical dispatch.

Exclusion Criteria:

* A subject who did not agree with this study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Time from 12-lead ECG device application starting to sending ECG result to hospital. | through study completion, an average of 2 month
  comparison of interval from the start of 12-lead ECG device application to complete of ECG result sending

SECONDARY OUTCOMES:
Usability of patchy-type wireless ECG device. | survey collecting through study completion an average of 2 month
  System Usability Scale survey of patchy-type wireless ECG device

CONTACTS AND LOCATIONS:
Overall Officials: tearim kim, doctoral, Principal Investigator — samsumg medical center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam, South Korea

REFERENCES:
- [Derived] Yoo S, Chang H, Kim T, Yoon H, Hwang SY, Shin TG, Sim MS, Jo IJ, Choi JH, Cha WC. Intervention in the Timeliness of Two Electrocardiography Types for Patients in the Emergency Department With Chest Pain: Randomized Controlled Trial. Interact J Med Res. 2022 Sep 13;11(2):e36335. doi: 10.2196/36335. PMID 36099010
- [Derived] Yoon S, Kim T, Roh T, Chang H, Hwang SY, Yoon H, Shin TG, Sim MS, Jo IJ, Cha WC. Twelve-Lead Electrocardiogram Acquisition With a Patchy-Type Wireless Device in Ambulance Transport: Simulation-Based Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Apr 1;9(4):e24142. doi: 10.2196/24142. PMID 33792550